CLINICAL TRIAL: NCT07256886
Title: Validation of the iCVS Model in Patients Admitted to the Intensive Care Unit: a Retrospective Study
Brief Title: Validation of the iCVS Model in Patients Admitted to the Intensive Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0289-25
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Shock
Keywords: shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with shock: Patients diagnosed with shock during ICU stay
- Patients without shock: Patients who were not diagnosed with shock during ICU stay

SUMMARY:
One of the significant challenges in the care of critically ill patients in the intensive care unit is the assessment of hemodynamically unstable patients (shock states). The treating team uses data such as heart rate, arterial blood pressure, physical examination findings, etc. to assess the patient's cardiac output, peripheral vascular resistance, filling pressures and volumes, and vascular tone. These assessments are essential to assess the cause of shock (cardiac cause, hypovolemia, sepsis, etc.), but in many situations they are not easy to perform and require extensive knowledge and experience. Assessing the hemodynamic status of a critically ill patient based on dynamic mechanical models may be a good option for more accurate assessment of complex patients. Such a model is, for example, the iCVS model: it is a relatively simple, mechanical-dynamic model that can be used to understand complex cardiovascular conditions. This model requires only age and weight as initial data, and as dynamic data the model requires only an arterial blood pressure (AR) curve and a central venous pressure (CVP) curve. The model is based on the shape of the above curves for the purpose of analyzing the cardiovascular status of the patient. The model is suitable for both adults and children, although most of the work to date has been among pediatric intensive care patients.

ELIGIBILITY:
Inclusion Criteria: The relevant experiment population are all patients over age 18 admitted to the ICU in Meir -

Exclusion Criteria: Missing data

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The relevant experiment population are all patients over age 18 admitted to the ICU in Meir. Research group: patients diagnosed with shock. Control group: patients not diagnosed with shock.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Optimization and validation of the ICVS model | 1 year
  The goal of this experiment is to perform an initial optimization and validation of the ICVS model with respect to the following metrics:
  * detection time before blood pressure drop
  * clinical shock classification.

IPD SHARING:
Plan to Share IPD: Undecided